CLINICAL TRIAL: NCT00892502
Title: Can Treatment With Bismuth Reduce Toxicity to Chemotherapy and Radiotherapy? A Clinical, Prospective, Randomized, Blinded Examination of Patients Suffering From Hematological Malignancies Treated With Intensive Chemotherapy and/or Radiotherapy.
Brief Title: Can Treatment With Bismuth Reduce Toxicity to Chemotherapy and Radiotherapy?
Acronym: Bismuth-PBH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007-007652-34
Record Dates: First submitted 2009-05-01; First posted 2009-05-04 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Hematological Diseases; Hematological Malignancies; Blood Diseases; Malignant Lymphoma; Leukemia; Multiple Myeloma
Keywords: haematology; haematological; hematology; hematological; malignancy; lymphoma; myeloma; leukemia; blood diseases; malignant; bismuth
MeSH Terms: conditions — Hematologic Diseases; Hematologic Neoplasms; Lymphoma; Leukemia; Multiple Myeloma; Neoplasms; Neoplasms, Plasma Cell | interventions — Bismuth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Bismuth tablets
  Interventions: Drug: Bismuth tablets
- 2 (Placebo Comparator): Placebo tablets, containing no active substance
  Interventions: Drug: Placebo tablets

INTERVENTIONS:
Drug: Bismuth tablets — 1000 mg x 2 for five days prior to chemotherapy/radiotherapy 500 mg x 2 for ten days during and after chemotherapy/radiotherapy
  Arms: 1
Drug: Placebo tablets — 1000 mg x 2 for five days prior to chemotherapy/radiotherapy 500 mg x 2 for ten days during and after chemotherapy/radiotherapy
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether treatment with Bismuth can reduce the toxicity of chemotherapy and radiotherapy in patients with malignant diseases of the blood.

ELIGIBILITY:
Inclusion Criteria:

* Patients of 18 years or over referred to the Department of Haematology L, Herlev Hospital, with a view to 'cytostatic'? treatment of or radiotherapy for haematological malignancy

Exclusion Criteria:

* Pregnant women and nursing mothers
* No informed consent from patient
* Known hyper sensitivity to bismuth or other tablet content
* Severe renal insufficiency with creatinin clearance below 25 ml/min.
* Patients receiving other treatment for protection of the mucous membrane except cryo treatment of the oral cavity (lumps of ice in the mouth)
* Other experimental treatment within past four weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-05; Primary Completion 2012-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
To evaluate a possible protective effect of bismuth on the mucous membranes during chemotherapy and radiotherapy | daily during treatment

SECONDARY OUTCOMES:
To identify the effect of bismuth on the regulation of metallothionein in tumour tissue and healthy tissue, respectively | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Per B Hansen, MD, Principal Investigator — Department of Haematology, Copenhagen University Hospital at Herlev
Locations (1):
- Department of Haematology L, Herlev Hospital, Herlev Ringvej 75, Herlev, Denmark